CLINICAL TRIAL: NCT00039494
Title: A Pilot and Phase II Study of OSI-774 and Temozolomide in Combination With Radiation Therapy in Glioblastoma Multiforme
Brief Title: Erlotinib and Temozolomide With Radiation Therapy in Treating Patients With Glioblastoma Multiforme or Other Brain Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00640; N0177; CDR0000069388; NCCTG-N0177; U10CA025224 (NIH)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Erlotinib Hydrochloride; Radiotherapy, Conformal; Temozolomide

ARMS (1):
- Treatment (erlotinib hydrochloride, radiation, temozolomide) (Experimental): Patients receive oral erlotinib once daily. After 1 week of erlotinib alone, patients also receive oral temozolomide once daily for 6 weeks and undergo concurrent radiotherapy 5 days a week for 6 weeks. After completion of radiotherapy, patients continue to receive erlotinib once daily alone in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after the completion of radiotherapy, patients also receive oral temozolomide once daily for 5 days. Temozolomide treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: erlotinib hydrochloride; Radiation: 3-dimensional conformal radiation therapy; Drug: temozolomide

INTERVENTIONS:
Drug: erlotinib hydrochloride — Given orally
  Other Names: CP-358,774; erlotinib; OSI-774
Radiation: 3-dimensional conformal radiation therapy
  Other Names: 3D conformal radiation therapy; 3D-CRT
Drug: temozolomide — Given orally
  Other Names: SCH 52365; Temodal; Temodar; TMZ

SUMMARY:
This pilot phase II trial is studying the side effects and best dose of erlotinib when given with temozolomide and radiation therapy and to see how well they work in treating patients with glioblastoma multiforme or other brain tumors. Radiation therapy uses high-energy x-rays to damage tumor cells. Erlotinib may interfere with the growth of tumor cells, slow the growth of the tumor, and make the tumor cells more sensitive to radiation therapy. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib and temozolomide with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PILOT STUDY OBJECTIVES:

I. Determine the maximum tolerated dose of erlotinib administered with temozolomide and radiotherapy in patients with glioblastoma multiforme or other grade 4 brain tumors who are currently on enzyme-inducing anticonvulsant (EIAC) therapy vs no EIAC therapy.

II. Determine the safety and tolerability of this regimen in these patients. III. Determine the toxic effects of this regimen in these patients. IV. Determine the efficacy of this regimen, in terms of 1-year survival, in these patients.

PHASE II OBJECTIVES:

I. Determine the response rate and time to progression in patients treated with this regimen.

II. Determine the 6-month progression-free survival of patients treated with this regimen.

III. Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation pilot study of erlotinib followed by a phase II study. Patients are stratified according to concurrent enzyme-inducing anticonvulsant drug use (yes vs no).

PILOT STUDY: Patients receive oral erlotinib once daily. After 1 week of erlotinib alone, patients also receive oral temozolomide once daily for 6 weeks and undergo concurrent radiotherapy 5 days a week for 6 weeks. After completion of radiotherapy, patients continue to receive erlotinib once daily alone in the absence of disease progression or unacceptable toxicity. Beginning 4 weeks after the completion of radiotherapy, patients also receive oral temozolomide once daily for 5 days. Temozolomide treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Once the MTD of erlotinib is determined, additional patients are treated with erlotinib at the MTD, temozolomide, and radiotherapy as above.

Patients are followed every 3 months for 5 years and then annually for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of 1 of the following:

  * Glioblastoma multiforme (grade 4 astrocytoma)
  * Gliosarcomas
  * Other grade 4 astrocytoma variants (e.g., giant cell)
* Must be enrolled at least 1 week, but no more than 4 weeks, after prior biopsy or surgery
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* At least 6 months
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* No inability to take oral medications
* No requirement for IV alimentation
* No active uncontrolled peptic ulcer disease
* No abnormalities of the cornea (e.g., dry eye syndrome or Sjögren's syndrome)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
* No abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)
* No prior allergy or intolerance to dacarbazine
* No other active malignancy requiring treatment
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior chemotherapy for any brain tumor
* No prior temozolomide
* No prior radiotherapy for any brain tumor
* No other concurrent investigational agents
* More than 21 days since prior major surgery (excluding neurosurgical biopsy or brain tumor resection)
* No prior surgical procedures affecting absorption
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2002-12; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Survival | At 52 weeks
Overall survival distribution | From start of study therapy to death due to any cause, up to 15 years
  The overall survival distribution will be estimated using the method of Kaplan-Meier. The success probability, i.e., 12-month survival percentage, will be estimated as the number of evaluable patients still alive at 366 days divided by the total number of evaluable patients followed for at least 366 days.

SECONDARY OUTCOMES:
Time-to-disease progression | From start of study therapy to documentation of disease progression, up to 15 years
  The time-to-progression distribution will be estimated using the Kaplan-Meier method.
Maximum toxicity grade, assessed by Common Terminology Criteria for Adverse Events (CTCAE) | Up to 15 years
  Frequency tables will be reviewed to determine toxicity patterns.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Brown, Principal Investigator — North Central Cancer Treatment Group
Locations (139):
- United States (139):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northeast Georgia Cancer Care LLC, Athens, Georgia
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Saint Anthony Memorial Hospital, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Saint Anthony Memorial Health Center, Michigan City, Indiana
  - McFarland Clinic, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Community Memorial Hospital, Missouri Valley, Iowa
  - Burgess Memorial Hospital, Onawa, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Harris, John Gilbert MD (UIA Investigator), Alexandria, Minnesota
  - Medini, Eitan MD (UIA Investigator), Alexandria, Minnesota
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Brainerd Medical Center Inc, Brainerd, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Etzell, Paul S MD (UIA Investigator), Fergus Falls, Minnesota
  - Swenson, Wade II, MD (UIA Investigator), Fergus Falls, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - Adult and Pediatric Urology PLLP, Sartell, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine of Bozeman, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Fremont Area Medical Center, Fremont, Nebraska
  - Bryan LGH Medical Center West, Lincoln, Nebraska
  - Bryan LGH Medical Center East, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - University of Virginia, Charlottesville, Virginia
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Brown PD, Krishnan S, Sarkaria JN, Wu W, Jaeckle KA, Uhm JH, Geoffroy FJ, Arusell R, Kitange G, Jenkins RB, Kugler JW, Morton RF, Rowland KM Jr, Mischel P, Yong WH, Scheithauer BW, Schiff D, Giannini C, Buckner JC; North Central Cancer Treatment Group Study N0177. Phase I/II trial of erlotinib and temozolomide with radiation therapy in the treatment of newly diagnosed glioblastoma multiforme: North Central Cancer Treatment Group Study N0177. J Clin Oncol. 2008 Dec 1;26(34):5603-9. doi: 10.1200/JCO.2008.18.0612. Epub 2008 Oct 27. PMID 18955445